CLINICAL TRIAL: NCT05796427
Title: Testing a Novel ADHD Engagement Intervention "START" to Improve Access to Treatment
Brief Title: Testing "SupporT for ADHD and Related Treatment" (START) for Families of Children With ADHD
Acronym: START
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Andrea Spencer, Vice Chair for Research in Psychiatry, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-5814
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-06

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- START Intervention (Experimental): Participants in the experimental group will be part of a 6-module weekly intervention where they will learn more about ADHD and its treatment.
  Interventions: Behavioral: SupporT for ADHD and Related Treatment
- Educational Brochure (No Intervention): Participants in the control group will receive an educational brochure by Children and Adults with Attention-Deficit/Hyperactivity Disorder (CHADD).

INTERVENTIONS:
Behavioral: SupporT for ADHD and Related Treatment — Intervention will include 6 modules typically taught over 6-7 weeks. Participants will have up to 3 months to complete the intervention. Modules will provide more knowledge on ADHD, discuss stigma around ADHD, address barriers in receiving care, encourage communication with physician and child, and empower caregivers. Overall, the goal being to improve engagement in ADHD treatment for newly diagnosed or unengaged families. This intervention is mostly targeted towards primary caregivers. However, the last module explicitly includes the child.
  Arms: START Intervention

SUMMARY:
The randomized control trial (RCT) study includes 2 aims; one being to test whether START increases access to treatment for ADHD. Investigators believe the intervention group will demonstrate improved treatment engagement and access to all treatments compared to controls. The second aim is to explore whether START leads to functional improvements across home, social and academic domains for the child and family. Investigators believe the intervention group will show better functioning including improved family and peer relationships and reduced parent stress compared to controls.

Before taking part in our study all participants will undergo a psychiatric evaluation. Eligible participants will be randomized to START while controls receive a pamphlet with ADHD information. Students and staff with related experience who are not mental health professionals will be trained to deliver START. START includes 6 modules, typically delivered over 6 sessions.

ELIGIBILITY:
Inclusion Criteria:

* The child is greater than or equal to 6 years old and less than or equal to 12 years old
* The child has a diagnosis of ADHD confirmed based on clinical psychiatric evaluation with an expert child psychiatrist on the study team (PI or Co-I)
* The diagnosis of ADHD is either new (defined as made for the first time by the study psychiatrist OR made for the first time within the prior 3 months by a medical or mental health provider) OR the child has been previously diagnosed but untreated either since diagnosis or for at least the prior 12 months. "Untreated" is defined as having received no therapeutic, medication, or school accommodations specifically for ADHD.
* They can understand and complete informed consent and study procedures in English.
* Children who have received treatment for other psychiatric conditions may be included if the treatment was specifically for a condition other than ADHD, to be confirmed by the study psychiatrist at enrollment.

Exclusion Criteria:

* Children with most comorbid (i.e., co-existing) psychiatric conditions with be included, but children with intellectual disability/cognitive impairment or psychotic symptoms will be excluded because these conditions would substantially change the focus of treatment
* Children under 6 and over 12 will be excluded because the intervention was specifically designed for school age children in this age group. Developmental, adolescents and preschoolers are considerably different than school age children and may require a different approach for engaging them and their parents in ADHD care. Children under 6 with ADHD symptoms may not yet be diagnosed and may not have the same treatment access or options as children 6 and over. Adolescents over 12 are more independent and an intervention may need to be more focused on the adolescent than our current intervention which is primarily parent focused.
* Children who were diagnosed over 3 months ago and already received treatment for ADHD will be excluded since our primary outcome is treatment engagement.
* Because this is an intervention only available in English at this time, participants who are not able to complete study procedures in English will be excluded.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Attention-deficit/hyperactivity disorder (ADHD) Treatment Utilization | 3 months
  Items from the National Survey of the Diagnosis and Treatment of ADHD and Tourette Syndrome (NS-DATA). Centers for Disease Control (CDC) survey used to evaluate treatment use among children with ADHD and Tourette syndrome.
Attention-deficit/hyperactivity disorder (ADHD) Symptoms and Functioning | 3 months
  Vanderbilt ADHD Diagnostic Rating Scale (VADRS). 55-item, parent-report questionnaire that assesses symptoms of ADHD and comorbidities as well as functional impairment in multiple domains (academics, family and peer relationships).

SECONDARY OUTCOMES:
Engagement Objectives | 3 months
  Attention-deficit/hyperactivity disorder (ADHD) Treatment Engagement Questionnaire. Developed by the PI for the pilot trial to assess engagement objectives directly corresponding to the conceptual model.
Parent ADHD Treatment Preferences | 3 months
  Attention-deficit/hyperactivity disorder (ADHD) Preference and Goal Instrument (PGI). Validated measure used in ADHD engagement studies that assesses parent perceptions of treatment feasibility, acceptability, and adverse effects for medication and therapy separately, as well as overall treatment goals.
Attention-deficit/hyperactivity disorder (ADHD) Knowledge | 3 months
  Attention-deficit/hyperactivity disorder (ADHD) Content Knowledge Questionnaire. 10-item parent quiz developed by the PI for the pilot trial and showing an increase in ADHD knowledge post-intervention.
Parent Activation | 3 months
  Parent-Patient Activation Measure (P-PAM). 13-item, parent-report measure adapted from the well-validated Patient Activation Measure (PAM) with acceptable reliability and validity.
Family Relationships | 3 months
  NIH Patient Reported Outcomes Measurement Information System (PROMIS) Pediatric Family Relationships Short Form. Created for the NIH PROMIS® using mixed methods, estimates the quality of the child's relationship with family in 8 items on a 5-point Likert scale with strong internal consistency and retest-reliability.
Parenting Stress | 3 months
  Parenting Stress Index-Short Form (PSI-SF) Brief, 36-item version of the full 120-item PSI, and one of the most common instruments used to measure parenting stress.
Social Risk | 3 months
  Child Healthwatch Vital Signs (food, housing, utilities)
Parent Self Stigma | 3 months
  Parents' Self Stigma Scale (PSSS)
  11-item scale assessing Parents' stigma
Parent Perceived Stigma | 3 months
  Parent Perceived Stigma of Services Seeking Scale (PPSSS)
  17-item scale assessing stigma toward seeking services for mental health resources
Child Education | 3 months
  Education Activation
  10-item scale assessing parents' involvement in child's education
ADHD School Services | 3 month
  Attention-deficit/hyperactivity disorder (ADHD) Preference and Goal Instrument (PGI)- School Services. Validated measure used in ADHD engagement studies that assesses school services.
ADHD Stages of Engagement Questionnaire | 3 months
  Survey identifies what stage of engagement the participant is in.

CONTACTS AND LOCATIONS:
Locations (1):
- Ann & Robert H. Lurie Children's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Visser SN, Danielson ML, Bitsko RH, Holbrook JR, Kogan MD, Ghandour RM, Perou R, Blumberg SJ. Trends in the parent-report of health care provider-diagnosed and medicated attention-deficit/hyperactivity disorder: United States, 2003-2011. J Am Acad Child Adolesc Psychiatry. 2014 Jan;53(1):34-46.e2. doi: 10.1016/j.jaac.2013.09.001. Epub 2013 Nov 21. PMID 24342384
- [Background] Cherkasova MV, Roy A, Molina BSG, Scott G, Weiss G, Barkley RA, Biederman J, Uchida M, Hinshaw SP, Owens EB, Hechtman L. Review: Adult Outcome as Seen Through Controlled Prospective Follow-up Studies of Children With Attention-Deficit/Hyperactivity Disorder Followed Into Adulthood. J Am Acad Child Adolesc Psychiatry. 2022 Mar;61(3):378-391. doi: 10.1016/j.jaac.2021.05.019. Epub 2021 Jun 8. PMID 34116167
- [Background] Shaw M, Hodgkins P, Caci H, Young S, Kahle J, Woods AG, Arnold LE. A systematic review and analysis of long-term outcomes in attention deficit hyperactivity disorder: effects of treatment and non-treatment. BMC Med. 2012 Sep 4;10:99. doi: 10.1186/1741-7015-10-99. PMID 22947230
- [Background] Coker TR, Elliott MN, Toomey SL, Schwebel DC, Cuccaro P, Tortolero Emery S, Davies SL, Visser SN, Schuster MA. Racial and Ethnic Disparities in ADHD Diagnosis and Treatment. Pediatrics. 2016 Sep;138(3):e20160407. doi: 10.1542/peds.2016-0407. Epub 2016 Aug 23. PMID 27553219
- [Background] Shi Y, Hunter Guevara LR, Dykhoff HJ, Sangaralingham LR, Phelan S, Zaccariello MJ, Warner DO. Racial Disparities in Diagnosis of Attention-Deficit/Hyperactivity Disorder in a US National Birth Cohort. JAMA Netw Open. 2021 Mar 1;4(3):e210321. doi: 10.1001/jamanetworkopen.2021.0321. PMID 33646315
- [Background] Geneva, WHO. Patient Engagement: Technical Series on Safer Primary Care. Published online 2016. Accessed January 7, 2022. https://apps.who.int/iris/bitstream/handle/10665/252269/9789241511629-eng.pdf
- [Background] Spencer AE, Sikov J, Loubeau JK, Zolli N, Baul T, Rabin M, Hasan S, Rosen K, Buonocore O, Lejeune J, Dayal R, Fortuna L, Borba C, Silverstein M. Six Stages of Engagement in ADHD Treatment Described by Diverse, Urban Parents. Pediatrics. 2021 Oct;148(4):e2021051261. doi: 10.1542/peds.2021-051261. Epub 2021 Sep 16. PMID 34531290
- [Background] Paidipati CP, Brawner B, Eiraldi R, Deatrick JA. Parent and Family Processes Related to ADHD Management in Ethnically Diverse Youth. J Am Psychiatr Nurses Assoc. 2017 Mar/Apr;23(2):90-112. doi: 10.1177/1078390316687023. Epub 2017 Jan 11. PMID 28076687
- [Background] Epstein JN, Kelleher KJ, Baum R, Brinkman WB, Peugh J, Gardner W, Lichtenstein P, Langberg J. Variability in ADHD care in community-based pediatrics. Pediatrics. 2014 Dec;134(6):1136-43. doi: 10.1542/peds.2014-1500. Epub 2014 Nov 3. PMID 25367532
- [Background] Brinkman WB, Epstein JN. Promoting productive interactions between parents and physicians in the treatment of children with attention-deficit/hyperactivity disorder. Expert Rev Neurother. 2011 Apr;11(4):579-88. doi: 10.1586/ern.10.151. PMID 21469930